CLINICAL TRIAL: NCT02586909
Title: A Long-Term, Open-Label Extension Study of the Safety and Tolerability of RVT-101 in Subjects With Alzheimer's Disease
Brief Title: 12-Month Open-Label Extension Study of Intepirdine (RVT-101) in Subjects With Alzheimer's Disease: MINDSET Extension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Intepirdine did't meet primary efficacy endpoints in lead-in study RVT-101-3001
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVT-101-3002
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; RVT-101; donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RVT-101 35 mg tablets (Experimental): once daily, oral tablets
  Interventions: Drug: RVT-101 35 mg tablets

INTERVENTIONS:
Drug: RVT-101 35 mg tablets — once daily, oral tablets

SUMMARY:
This 12-month open-label study will provide further information regarding the long-term safety and tolerability of intepirdine (RVT-101) for subjects with Alzheimer's disease who have completed the double-blind, placebo-controlled, lead-in study RVT-101-3001 (double-blind study).

DETAILED DESCRIPTION:
This 12-month open-label study will provide further information regarding the long-term safety and tolerability of intepirdine (RVT-101) for subjects with Alzheimer's disease who have completed the double-blind, placebo-controlled, lead-in study RVT-101-3001. Various background therapies, including acetylcholinesterase inhibitors and memantine, will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Completed last on-treatment visit of the lead-in study RVT-101-3001

Exclusion Criteria:

* Any clinically relevant concomitant disease, which, in the opinion of the investigator, makes the subject unsuitable for inclusion in the study.

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1099 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences, Inc., Vice President, Clinical Research
Locations (168):
- United States (52):
  - US112, Phoenix, Arizona
  - US220, Tucson, Arizona
  - US096, Rancho Mirage, California
  - US195, Santa Ana, California
  - US016, Simi Valley, California
  - US106, Temecula, California
  - US179, Hamden, Connecticut
  - US171, Norwich, Connecticut
  - US088, Atlantis, Florida
  - US007, Brooksville, Florida
  - US002, Hallandale, Florida
  - US140, Hialeah, Florida
  - US216, Miami, Florida
  - US110, Miami, Florida
  - US172, North Palm Beach, Florida
  - US003, Orlando, Florida
  - US256, Pensacola, Florida
  - US037, Tampa, Florida
  - US042, Tampa, Florida
  - US004, The Villages, Florida
  - US048, Atlanta, Georgia
  - US046, Atlanta, Georgia
  - US217, Columbus, Georgia
  - US111, Baton Rouge, Louisiana
  - US095, Shreveport, Louisiana
  - US116, Newton, Massachusetts
  - US174, Quincy, Massachusetts
  - US144, Hattiesburg, Mississippi
  - US094, Las Vegas, Nevada
  - US135, Berlin, New Jersey
  - US197, Lawrenceville, New Jersey
  - US215, Mount Arlington, New Jersey
  - US057, Paterson, New Jersey
  - US209, Toms River, New Jersey
  - US036, West Long Branch, New Jersey
  - US001, Albany, New York
  - US049, Brooklyn, New York
  - US097, New Hyde Park, New York
  - US044, New York, New York
  - US150, Chapel Hill, North Carolina
  - US185, Charlotte, North Carolina
  - US008, Cincinnati, Ohio
  - US113, Cleveland, Ohio
  - US119, Shaker Heights, Ohio
  - US134, Portland, Oregon
  - US169, Media, Pennsylvania
  - US162, Plains, Pennsylvania
  - US148, Willow Grove, Pennsylvania
  - US043, San Antonio, Texas
  - US143, Orem, Utah
  - US149, Charlottesville, Virginia
  - US170, Spokane, Washington
- Argentina (17):
  - AR130, La Plata, Buenos Aires
  - AR101, Buenos Aires
  - AR060, Buenos Aires
  - AR084, Ciudad Autonoma de Buenos Aire
  - AR027, Ciudad Autonoma de Buenos Aire
  - AR012, Ciudad Autonoma de Buenos Aire
  - AR160, Ciudad Autonoma de Buenos Aire
  - AR028, Ciudad Autonoma de Buenos Aire
  - AR035, Ciudad Autonoma de Buenos Aire
  - AR040, Ciudad Autónoma de Buenos Aire
  - AR081, Ciudad Autónoma de Buenos Aire
  - AR051, Córdoba
  - AR137, Córdoba
  - AR126, Córdoba
  - AR210, Mendoza
  - AR219, Mendoza
  - AR059, Santiago del Estero
- Australia (4):
  - AU227, Caulfield
  - AU032, Heidelberg West
  - AU011, Hornsby
  - AU138, West Perth
- Bulgaria (3):
  - BU125, Rousse
  - BU131, Sofia
  - BU073, Varna
- Canada (7):
  - CA054, Kelowna, British Columbia
  - CA188, Kelowna, British Columbia
  - CA186, Penticton, British Columbia
  - CA141, West Vancouver, British Columbia
  - CA147, Newmarket, Ontario
  - CA196, North York, Ontario
  - CA236, Gatineau, Quebec
- Chile (4):
  - CH212, Antofagasta, Antofagasta
  - CH061, Santiago, Santiago Metropolitan
  - CH075, Santiago, Santiago Metropolitan
  - CH076, Santiago, Santiago Metropolitan
- Croatia (3):
  - CR069, Zagreb
  - CR122, Zagreb
  - CR070, Zagreb
- Czechia (5):
  - CZE128, Prague
  - CZE207, Prague
  - CZE132, Prague
  - CZE129, Prague
  - CZE161, Rychnov nad Kněžnou
- France (4):
  - FR231, Lille
  - FR182, Marseille
  - FR221, Paris
  - FR202, Villeurbanne
- Germany (12):
  - GE206, Bad Homburg
  - GE091, Berlin
  - GE071, Berlin
  - GE139, Berlin
  - GE230, Cologne
  - GE252, Ellwangen
  - GE180, Leipzig
  - GE228, Mannheim
  - GE017, München
  - GE157, Nuremberg
  - GE098, Ulm
  - GE251, Westerstede
- Italy (9):
  - IT053, Brescia
  - IT124, Cefalù
  - IT030, Pavia
  - IT103, Perugia
  - IT072, Roma
  - IT029, Roma
  - IT183, Rome
  - IT175, Rome
  - IT085, Torino
- Poland (8):
  - PO013, Bialystok
  - PO024, Bydgoszcz
  - PO010, Bydgoszcz
  - PO107, Katowice
  - PO092, Katowice
  - PO009, Poznan
  - PO014, Szczecin
  - PO074, Warsaw
- Serbia (6):
  - SE164, Belgrade
  - SE193, Belgrade
  - SE090, Belgrade
  - SE155, Kragujevac
  - SE031, Novi Kneževac
  - SE165, Vršac
- Singapore (2):
  - SI052, Singapore
  - SI026, Singapore
- Slovakia (4):
  - SL056, Banská Bystrica
  - SL200, Dubnica nad Váhom
  - SL078, Krompachy
  - SL077, Svidník
- South Korea (3):
  - SK066, Busan
  - SK067, Seoul
  - SK190, Seoul
- Spain (8):
  - SP249, Alicante
  - SP176, Barcelona
  - SP022, Barcelona
  - SP021, Barcelona
  - SP250, Barcelona
  - SP184, Barcelona
  - SP222, Getxo
  - SP194, San Sebastián
- TA121, Taoyuan District, Taiwan
- United Kingdom (16):
  - UK063, Bath
  - UK038, Blackpool
  - UK233, Cambridge
  - UK033, Carnoch
  - UK211, Epping
  - UK234, Guildford
  - UK055, Leeds
  - UK039, London
  - UK034, Manchester
  - UK087, Oxford
  - UK235, Plymouth
  - UK100, Sheffield
  - UK064, Southampton
  - UK152, Southampton
  - UK153, Swindon
  - UK154, Warrington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RVT-101 35 mg Tablets
Started | 1099
Completed | 151
Not Completed | 948

BASELINE CHARACTERISTICS:
Arm/Group | RVT-101 35 mg Tablets
Number analyzed (Participants) | 1099
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 158
  >=65 years | 941
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 676
  Male | 423
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 193
  Not Hispanic or Latino | 897
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 44
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 1022
  More than one race | 0
  Unknown or Not Reported | 16
Region of Enrollment [Number; unit: participants]
  Argentina | 103
  Singapore | 16
  United States | 281
  Czechia | 53
  United Kingdom | 164
  Spain | 65
  Canada | 37
  South Korea | 9
  Taiwan | 16
  Poland | 47
  Italy | 61
  Slovakia | 42
  Australia | 31
  Bulgaria | 7
  Chile | 48
  France | 13
  Serbia | 21
  Germany | 55
  Croatia | 30
Height [Mean (Standard Deviation); unit: cm] | 163.3 (9.86)
Weight [Mean (Standard Deviation); unit: kg] | 71.08 (14.490)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.59 (4.653)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events (AEs) and or Reported Changes in Physical Examinations, Vital Signs Measurements, Electrocardiograms (ECGs), Routine Laboratory Assessments
Description: The primary outcome measure is to study the safety of Intepridine (RVT-101) by determining the incidence of AEs, changes in physical examinations, vital signs measurements, ECGs and clinical laboratory assessments
Time Frame: Baseline to 12 months or Early Termination
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-101 35 mg Tablets
Number analyzed (Participants) | 1099
Participants
  Subjects with at least one on-treatment AE | 549
  Subjects with no on-Treatment AE | 550

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | RVT-101 35 mg Tablets
All-Cause Mortality (participants affected / at risk) | 10/1099
Serious Adverse Events (participants affected / at risk) | 87/1099
Other Adverse Events (participants affected / at risk) | 526/1099
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RVT-101 35 mg Tablets (N=1099)
Pneumonia (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Appendicitis perforated (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 5
Accidental overdose (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 2
Sinus node dysfunction (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Heart valve stenosis (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastritis erosive (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Pancreatic cyst (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dementia of the Alzheimer's type, with delirium (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Deep vein thrombosis (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Hypothermia (General disorders) | 1
Sudden death (General disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Full blood count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Cervix disorder (Reproductive system and breast disorders) | 1
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RVT-101 35 mg Tablets (N=1099)
Anaemia (Blood and lymphatic system disorders) | 9
Eosinophilia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutrophilia (Blood and lymphatic system disorders) | 2
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 3
Sinus arrhythmia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 2
Cerumen impaction (Ear and labyrinth disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 7
Hypothyroidism (Endocrine disorders) | 3
Thyroid mass (Endocrine disorders) | 1
Angle closure glaucoma (Eye disorders) | 1
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 8
Dry eye (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Ocular rosacea (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Anal fissure (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 17
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Faeces soft (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 3
Hiatus hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Oral contusion (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Umbilical hernia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Chest pain (General disorders) | 2
Facial pain (General disorders) | 1
Fat necrosis (General disorders) | 1
Fatigue (General disorders) | 4
Feeling cold (General disorders) | 1
Gait disturbance (General disorders) | 6
Gravitational oedema (General disorders) | 1
Hyperthermia (General disorders) | 1
Influenza like illness (General disorders) | 2
Non-cardiac chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 1
Thirst (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 3
Bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 12
Bronchitis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 6
Gastroenteritis viral (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Hordeolum (Infections and infestations) | 1
Infected bite (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 1
Influenza (Infections and infestations) | 7
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 6
Lyme disease (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 23
Onychomycosis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Postoperative wound infection (Infections and infestations) | 1
Pyuria (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Root canal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 45
Urinary tract infection bacterial (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Asbestosis (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 10
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Dose calculation error (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 51
Forearm fracture (Injury, poisoning and procedural complications) | 1
Frostbite (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 3
Head injury (Injury, poisoning and procedural complications) | 5
Heat stroke (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 6
Skin injury (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2
Splinter (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 3
Ulna fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Wound secretion (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 6
Blood electrolytes abnormal (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood potassium increased (Investigations) | 2
Blood pressure increased (Investigations) | 4
Blood urea increased (Investigations) | 3
Blood urine present (Investigations) | 2
Creatinine renal clearance decreased (Investigations) | 15
Crystal urine (Investigations) | 1
Crystal urine present (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 14
Glomerular filtration rate decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Liver function test increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 8
Mammogram abnormal (Investigations) | 1
Monocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Neutrophil count increased (Investigations) | 3
Platelet count decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Red blood cell count increased (Investigations) | 1
Red blood cells urine (Investigations) | 1
Transaminases increased (Investigations) | 1
Urine analysis abnormal (Investigations) | 4
Urine leukocyte esterase (Investigations) | 1
Weight decreased (Investigations) | 7
Weight increased (Investigations) | 5
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Food craving (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Underweight (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 22
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Apraxia (Nervous system disorders) | 1
Areflexia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Bradykinesia (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Cervicobrachial syndrome (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 4
Decreased vibratory sense (Nervous system disorders) | 3
Dementia Alzheimer's type (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 17
Dizziness postural (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspraxia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Facial paralysis (Nervous system disorders) | 1
Gait apraxia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 17
Hypertonia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Parkinsonian gait (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 3
Postural tremor (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 6
Tension headache (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 4
Abnormal behaviour (Psychiatric disorders) | 5
Abnormal dreams (Psychiatric disorders) | 2
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 8
Agitation (Psychiatric disorders) | 17
Anxiety (Psychiatric disorders) | 16
Confusional state (Psychiatric disorders) | 7
Delirium (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 7
Depressed mood (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 14
Disorientation (Psychiatric disorders) | 3
Dysphemia (Psychiatric disorders) | 1
Encopresis (Psychiatric disorders) | 1
Enuresis (Psychiatric disorders) | 1
Frustration tolerance decreased (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 4
Hallucination, olfactory (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 8
Irritability (Psychiatric disorders) | 11
Libido decreased (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 2
Mood swings (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Neuropsychiatric symptoms (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 2
Paranoia (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 3
Sleep disorder (Psychiatric disorders) | 5
Suicidal ideation (Psychiatric disorders) | 5
Suspiciousness (Psychiatric disorders) | 1
Tearfulness (Psychiatric disorders) | 2
Calculus bladder (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 4
Hypertonic bladder (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 4
Polyuria (Renal and urinary disorders) | 2
Renal cyst (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Ureterolithiasis (Renal and urinary disorders) | 3
Urethral fistula (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 12
Urinary retention (Renal and urinary disorders) | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Breast haematoma (Reproductive system and breast disorders) | 1
Cervix disorder (Reproductive system and breast disorders) | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 1
Prostatomegaly (Reproductive system and breast disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2
Macule (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Rash generalised (Skin and subcutaneous tissue disorders) | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Blood pressure fluctuation (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 3
Orthostatic hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 1
Peripheral venous disease (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02586909/Prot_SAP_000.pdf